CLINICAL TRIAL: NCT04250220
Title: eHealth-based Bavarian Alternative Detection of Atrial Fibrillation: A Randomized Controlled Trial (eBRAVE-AF)
Acronym: eBRAVE-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LMU Klinikum (Other)
Collaborators: Preventicus GmbH (Industry); Versicherungskammer Bayern (Unknown)
Responsible Party: Principal Investigator, Axel Bauer, Prof. Dr., LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-779
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): e-health-based strategy
  Interventions: Diagnostic Test: e-Health based strategy: PPG-based screening using a smartphone and ECG patch
- control group (No Intervention): symptom based AF-screening

INTERVENTIONS:
Diagnostic Test: e-Health based strategy: PPG-based screening using a smartphone and ECG patch — PPG-analysis via Smartphone-App (Preventicus Heart Beats) and ECG patch
  Arms: intervention group

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia in western countries and causes of up to one quarter of ischemic strokes. The randomized eHealth-based Bavarian Alternative Detection of Atrial Fibrillation study (eBRAVE-AF) tests the efficacy of an e-health based strategy for the detection of AF. The e-health-based strategy consists of a smartphone-based photophlethysmographic (PPG) screening and an ECG-based validation.

ELIGIBILITY:
Inclusion Criteria:

* policy holders of a large health insurance company
* age ≥50 years
* CHA2DS2-VASc ≥1 (females ≥2)

Exclusion Criteria:

* atrial fibrillation
* oral anticoagulation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with newly diagnosed atrial fibrillation within six months with prescription of oral anticoagulation | 6 months

SECONDARY OUTCOMES:
Number of participants with newly diagnosed atrial fibrillation | 6 months
Number of participants with newly prescribed oral anticoagulation | 6 months
Number of participants with stroke | 6 months
Number of participants with thromboembolic events | 6 months

OTHER OUTCOMES:
Number of participants with TIMI major bleeding | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Axel Bauer, MD, Principal Investigator — LMU Klinikum
Locations (1):
- Klinikum der Universität München, München, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizas KD, Freyer L, Sappler N, von Stulpnagel L, Spielbichler P, Krasniqi A, Schreinlechner M, Wenner FN, Theurl F, Behroz A, Eiffener E, Klemm MP, Schneidewind A, Zens M, Dolejsi T, Mansmann U, Massberg S, Bauer A. Smartphone-based screening for atrial fibrillation: a pragmatic randomized clinical trial. Nat Med. 2022 Sep;28(9):1823-1830. doi: 10.1038/s41591-022-01979-w. Epub 2022 Aug 28. PMID 36031651
- [Derived] Freyer L, von Stulpnagel L, Spielbichler P, Sappler N, Wenner F, Schreinlechner M, Krasniqi A, Behroz A, Eiffener E, Zens M, Dolejsi T, Massberg S, Rizas KD, Bauer A. Rationale and design of a digital trial using smartphones to detect subclinical atrial fibrillation in a population at risk: The eHealth-based bavarian alternative detection of Atrial Fibrillation (eBRAVE-AF) trial. Am Heart J. 2021 Nov;241:26-34. doi: 10.1016/j.ahj.2021.06.008. Epub 2021 Jul 9. PMID 34252387